CLINICAL TRIAL: NCT03242837
Title: Psychobiological Evaluation of the Army Resilience Training
Acronym: OpPHX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Military Academy at ETH Zurich (Other Government)
Collaborators: Swiss Armed Forces (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Project ID 2017-00841
Record Dates: First submitted 2017-07-26; First posted 2017-08-08 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Psychological Stress; Psychological Adaptation
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Army Resilience Training (Experimental): Resilience training: four training sessions of 90 minutes each (in week 3, 5, 6 and 7 of military training), in classroom, psychoeducational inputs on stress management and resilience related topics, cognitive behavioral interventions and moderated exercises
  Interventions: Behavioral: Army Resilience Training
- Diversity Management Training (Active Comparator): Diversity Management: four training sessions of 90 minutes each (in week 3, 5, 6 and 7 of military training), classroom, psychoeducational inputs on social awareness and exercises
  Interventions: Other: Diversity Management Training

INTERVENTIONS:
Behavioral: Army Resilience Training — The Army Resilience Training consists four training sessions of 90 minutes each. Participants learn to reflect their stress management (including thinking, emotions, behavioral consequences; coping strategies) and build resilience using specific strategies.
  Other Names: Resilience Training
  Arms: Army Resilience Training
Other: Diversity Management Training — Diversity Management Training consists four training sessions of 90 minutes each. Participants learn about diversity and social awareness reflecting different situations and settings.
  Other Names: Diversity Management
  Arms: Diversity Management Training

SUMMARY:
This study evaluates the influence of a resilience training on psychobiological factors which are related to stress and resilience in young healthy male cadets. Half of participants will join in the resilience training, while the other half take part in a control-training (diversity management training).

DETAILED DESCRIPTION:
The resilience training (Army Resilience Training / ART) is a stress prevention program based on well established methods from Cognitive Behavioral Therapy (CBT) and Positive Psychology adapted for the needs of Swiss Armed Forces. ART is designed for healthy subjects to learn how to get over strain.

Diversity management training (DMT) aims to promote social skills and acts as control condition. DMT is part of the military training but not mandatory for the study population.

ELIGIBILITY:
Inclusion Criteria:

* military cadets of the Swiss Army Infantry Officers School Inf OS 10-1/17

Exclusion Criteria:

* no

Ages: 18 Years to 28 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-08-17 (Actual)

PRIMARY OUTCOMES:
Change in heart rate variability (HRV) | Weeks 2 (baseline) and 9 of the military training
  Change is the difference from HRV at baseline (week 2) and after resilience training (intervention) in week 9
Area under the curve (AUC) with respect to changes of salivary cortisol titer | Weeks 2 and 9 of the military training
  During stress exposure; six saliva samples will be taken and analyzed for cortisol reactivity.
Change of Testosterone Levels | Weeks 2 and 9 of the military training
  During stress exposure; four saliva samples will be taken and analyzed for testosterone levels.

SECONDARY OUTCOMES:
Intensity of acute psychological stress | Weeks 2, 9 and 12 of the military training
  Perceived stress intensity measured by Visual Analogue Scale
Affect of acute psychological stress | Weeks 2, 9 and 12 of the military training
  Perceived stress measured by Positive Negative Affect
Stress Appraisal | Weeks 2, 9 and 12 of the military training
  Perceived stress appraisal measured by Primary and Secondary Appraisal

OTHER OUTCOMES:
Resilience | Weeks 1 and 15 of the military training and follow-up (+7 months)
  Resilience measured by following questionnaire: Brief Resilience Scale
Psychological Resistance | Weeks 1 and 15 of the military training and follow-up (+7 months)
  Psychological Resistance measured by following questionnaire: Resilience Scale RS-11
Perceived Stress | BWeeks 1 and 15 of the military training and follow-up (+7 months)
  Stress management measured by following questionnaire: Perceived Stress Questionnaire
Stress Reactivity | BWeeks 1 and 15 of the military training and follow-up (+7 months)
  Stress management measured by following questionnaire: Stress Reactivity Scale
Coping Strategies | Weeks 1 and 15 of the military training and follow-up (+7 months)
  Stress management measured by following questionnaire: Coping Inventory for Stressful Situations
Cognitive Emotion Regulation | Weeks 1 and 15 of the military training and follow-up (+7 months)
  Stress management measured by following questionnaire: Cognitive Emotion Regulation Questionnaire
Personality | Weeks 1 and 15 of the military training and follow-up (+7 months)
  Personality measured by following questionnaire: NEO-Five Factor Inventory
Dark Triad | Weeks 1 and 15 of the military training and follow-up (+7 months)
  Dark Triad measured by following questionnaire: Dark Triad / Dirty Dozen
Self-Esteem | Weeks 1 and 15 of the military training and follow-up (+7 months)
  Self-Esteem measured by following questionnaire: Rosenberg Self Esteem Scale
Optimism | Weeks 1 and 15 of the military training and follow-up (+7 months)
  Optimism measured by following questionnaire: Life Orientation Test
Social Support | Weeks 1 and 15 of the military training and follow-up (+7 months)
  Social Support measured by following questionnaire: Berlin Social Support Scales
Health | Weeks 1 and 15 of the military training and follow-up (+7 months)
  Health measured by following questionnaire: Maastricht Vital Exhaustion Questionnaire
Sleep | Weeks 1 and 15 of the military training and follow-up (+7 months)
  Sleep measured by following questionnaire: Pittsburgh Sleep Quality Index
Leadership | Follow-up (+7 months)
  Leadership measured by following questionnaire: Leader Member Exchange

CONTACTS AND LOCATIONS:
Overall Officials: Hubert Annen, PhD, Principal Investigator — Military Academy at ETH Zurich
Locations (1):
- Swiss Military Caserne, Liestal, Basel-Landschaft, Switzerland

IPD SHARING:
Plan to Share IPD: No